CLINICAL TRIAL: NCT06977165
Title: Investigating the Impact of Sepsis Phenotypes on Antibiotic Treatment in Patients With Severe Pneumonia and Sepsis: a Prospective Observational Cohort Study
Brief Title: Investigating the Impact of Sepsis Phenotypes on Antibiotic Treatment in Patients With Severe Pneumonia and Sepsis
Acronym: SIPRES
Status: Not yet recruiting | Type: Observational
Sponsor: University of Manchester (Other)
Responsible Party: Sponsor
Other Study IDs: R131285; NIHR304654 (Other Grant/Funding Number: National Institute for Health and Care Research)
Record Dates: First submitted 2025-05-08; First posted 2025-05-18 (Actual); Last update posted 2025-05-18 (Actual); Status verified 2025-05

CONDITIONS: Respiration Disorders; Respiratory Failure; Sepsis; Infection in ICU; Pneumonia
Keywords: sepsis; pneumonia; therapeutic drug monitoring; beta-lactam antibiotics; piperacillin-tazobactam
MeSH Terms: conditions — Respiration Disorders; Respiratory Insufficiency; Sepsis; Pneumonia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood and sputum
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Antibiotic quantification — Piperacillin/tazobactam quantification using liquid chromatography-tandem mass spectrometry

SUMMARY:
Aim of the research: To find out why antibiotics work differently in certain patients with severe pneumonia and sepsis.

Background: Individuals can become very unwell from pneumonia, sometimes requiring admission to hospital or even the intensive care unit (ICU). In some cases, pneumonia can lead to a condition called sepsis, which can be deadly if not treated quickly. In the UK, approximately 30,000 patients die from pneumonia every year. Clinicians use antibiotic injections to treat life-threatening infections such as severe pneumonia. After being injected into the bloodstream, antibiotics quickly spread throughout the body, attacking the infection. Antibiotics are eventually broken down and removed from the body by the kidneys and other organs. However, antibiotics fail to achieve the same consistent result for every patient. This may be to do with the way the antibiotics travel through and are removed from the body, leading to different antibiotic levels in the blood at any one time. Low antibiotic levels can result in worse outcomes and antibiotic resistance. Patients can be grouped based on how their immune system reacts to infections. The SIPRES Study aims to explore if these previously described groups explain the difference in antibiotic levels in patients with severe pneumonia and sepsis.

Procedures: We will study how adult patients with severe pneumonia respond when treated with the most commonly used antibiotic in the ICU called piperacillin/tazobactam. Alongside information on how quickly patients get better and how long they need to stay in hospital or in ICU, we will collect blood samples to measure antibiotic levels and assess each patient's immune system at two time points during their treatment. This will allow us to measure antibiotic levels in blood at different times and group patients based on their immune system reaction to infection. We will describe the range of antibiotic levels seen in the different immune system reaction groups using mathematical and statistical models.

Patient involvement: We are working closely with people who have experienced severe pneumonia and will work with two patient partners and a patient advisory group to help shape this research. Patient contributors have already shaped the development of the funding application and identified important study outcomes. Patients we have spoken to are concerned over the appropriate dosing of antibiotics and appreciate the need for improved and precise approaches to treating severe infections. Moving forward, patient partners will help finalise the protocol, develop patient and public facing materials, provide their perspective on the study results and shape plans to share the outcomes of the study more broadly.

Potential impact: The SIPRES Study will help identify a group of patients at risk of low antibiotic levels in blood, who are less likely to improve with treatment and more likely to develop antibiotic resistance. Mathematical models that can help clinicians personalise antibiotic dosing for each critically ill patient with severe pneumonia will be developed. Findings have the potential to limit the development of antibiotic resistance and help patients survive and get better faster so that they can return to their normal daily lives. Individualised dosing for patients with low antibiotic levels, as opposed to 'one size fits all' prescribing, also has the potential to more efficiently allocate scarce resources to those who will benefit the most.

ELIGIBILITY:
Inclusion Criteria:

* age ≥ 18 years;
* admitted to intensive care and receiving at least one-organ supportive care;
* treated for presumed or confirmed lower respiratory infection;
* receiving or about to receive piperacillin/tazobactam as part of standard clinical care;
* valid informed consent or enrolment through deferred consent pathway appropriate.

Exclusion Criteria:

* unlikely to survive 24 hours as judged by the treating physician;
* study antimicrobial started more than 24 hours prior.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hospitalised critically ill patients admitted to the intensive care unit
Sampling Method: Non-Probability Sample
Enrollment: 119 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
Serum concentrations of antimicrobial | Day 0 ± Day 3-5
  The primary outcome of serum concentrations of antimicrobials was chosen to assess the profile of medication processing in the body between the groups of interest. Multiple blood samples are taken over the space of one dosing interval (most often 6-8 hours for piperacillin/tazobactam), which allows the calculation of an area under the concentration curve over time. For participants who remain in ICU at Visit 2 (Day 3-5) and are still receiving antimicrobials, a second sampling episode will occur. Those discharged from ICU prior will undergo only a single sampling period.

SECONDARY OUTCOMES:
Baseline Sequential Organ Failure Assessment score (SOFA) | Day 0
  SOFA score at baseline
Change in SOFA score | From Day 0 to Day 3-5
  Difference between aggregate SOFA scores
All-cause mortality | At Day 28
  Death censored at Day 28
Days alive and out of hospital | At Day 28
  Defined as the number of days not in hospital at Day 28
Hospital and ICU length of stay | At Day 28
  Number of days in hospital/ICU
Clinical cure | At Day 28
  Defined as the completion of antibiotic treatment course (on or prior to Day 28) without recommencement of antibiotic therapy within 48 hours of cessation
Microbiological cure | At Day 28
  Defined as at least two negative cultures following proven bacterial infection and no new positive cultures at Day 28
Duration of primary course of antimicrobial treatment | At Day 28
  Number of days of treatment with antimicrobial from baseline
Isolated pathogens | At Day 28
  Proportion of participants with isolated pathogens
Emergence of resistant organisms | At Day 28
  Any organism resistant to antimicrobials identified through culture from any source (blood, urine, sputum, stool)
Therapeutic target attainment | At Day 0 ± Day 3-5
  100% fraction of the time (fT) above the minimal inhibitory concentration [MIC] 100% fraction of the time (fT) above four times the minimal inhibitory concentration [4xMIC] Assessed for Pseudomonas aeruginosa according to latest EUCAST ECOFF breakpoints at time of analysis
Immune signature | At Day 0 ± Day 3-5
  Phenotype category according to Davenport and Sinha classification
Safety and toxicity outcomes | At Day 28
  Any serious adverse events reported during the study period

CONTACTS AND LOCATIONS:
Locations (1):
- The University of Manchester, Manchester, Lancashire, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
The following anonymised data will be shared on an online accessible repository in line with Findability, Accessibility, Interoperability, and Reuse (FAIR) principles:
  * Baseline clinical characteristics without identifiable data
  * Outcome data
  * Pharmacokinetic data
  * Transcriptomic data
  * Immune cytokine data
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Beginning one year after publication and indefinitely
Access Criteria: A limited anonymised dataset will be shared openly, allowing secondary analyses; more detailed IPD may be shared with researchers upon reasonable request.